CLINICAL TRIAL: NCT05724355
Title: Dalpiciclib Combined With Camrelizumab for PD-1 Inhibitor Refractory R/M NPC
Brief Title: CDK4/6 Inhibitor Plus Camrelizumab for PD-1 Inhibitor Refractory R/M NPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Chief physician, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2022-CDK46
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dalpiciclib plus Camrelizumab (Experimental)
  Interventions: Drug: Dalpiciclib Isetionate Tablets, Camrelizumab

INTERVENTIONS:
Drug: Dalpiciclib Isetionate Tablets, Camrelizumab — Dalpiciclib, D1-21, po, 150mg, qd, Q4W. Camrelizumab, iv, 200mg, D1, Q3W.

SUMMARY:
Because most patients with R/M NPC have received long-term maintenance of immunotherapy at the time of initial treatment and the first-line treatment, there are a large number of PD-1 inhibitor refractory patients. How to deal with the ICIs resistance is an urgent problem in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Had histopathologically confirmed nonkeratinizing recurrent/metastatic NPC.
2. ECOG performance status of 0 or 1.
3. Progression after previous treatment with platinum-based dual-drug chemotherapy.
4. Progression after previous treatment with PD-1 inhibitors.
5. Experieced at least 1 line systemic therapy.
6. Subjects enrolled must have measurable lesion(s) according to response evaluation criteria in solid (RECIST) v1.1.
7. Adequate organ function assessed by laboratory parameters during the screening period.
8. Life expectancy more than 12 weeks.
9. Able to understand and sign an informed consent form (ICF).
10. Able to swallow the pill.

Exclusion Criteria:

1. Recurrent lesions suitable for radical treatment (radiotherapy or surgery).
2. Previous treatment over 3 lines.
3. Prior use of CDK4/6 inhibitors.
4. Patients with other malignancies.
5. Patients with known or suspected autoimmune diseases including dementia and seizures.
6. Multiple factors affecting the absorption of oral medications (e.g., dysphagia, chronic diarrhea, and bowel obstruction).
7. An excessive dose of glucocorticoids given within 4 weeks before enrollment.
8. Complications requiring long-term use of immunosuppressive drugs or systemic or local use of immunosuppressive-dose corticosteroids.
9. Patients with active pulmonary tuberculosis (TB) receiving anti-TB treatment or who have received anti-TB treatment within 1 year prior to screening.
10. HIV positive; HBsAg positive and HBV DNA copy number positive (quantitative detection ≥ 1000 cps/ml); chronic hepatitis C with blood screening positive (HCV antibody positive).
11. Any anti-infective vaccines such as influenza vaccine, varicella vaccine, etc., within 4 weeks before enrollment.
12. Women of childbearing age with a positive pregnancy test and lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 year
  Objective response rate is the rate of patients achieving complete response or partial response for a certain period of time after intervention.

SECONDARY OUTCOMES:
Median progression-free survival (PFS) | 1 year
  Progression-free survival is defined as the time to the date of death of any cause or the first progress at any site, censored on the last date of tumor evaluation if no progress has happened.
Median overall survival (OS) | 3 years
  Overall survival is defined as the time to the date of death of any cause, censored on the last date of known survival if no death has happened.
Duration of response (DoR) | 1 year
  Defined as the time from first documentation of objective response to radiological disease progression
Disease control rate (DCR) | 1 year
  Disease control rate is the rate of patients achieving complete response, partial response or stable disease
Incidence of adverse events | 1 year
  NCI-CTCAE 5.0 standard is adopted.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China